CLINICAL TRIAL: NCT01821040
Title: A Randomised, Multi-centre, Double-blind, Active-controlled, Parallel Group Study to Assess the Efficacy and Safety of Modified Release Prednisone (Lodotra®) Compared to Immediate Release Prednisone (Prednisone IR) in Subjects Suffering From Polymyalgia Rheumatica (PMR).
Brief Title: A Study Assessing the Efficacy and Safety of Lodotra® Compared to Prednisone IR in Subjects Suffering From PMR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOD3501; 2011-002353-57 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-03-29 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia rheumatica; PMR; Modified release prednisone
MeSH Terms: conditions — Polymyalgia Rheumatica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lodotra® (Experimental): Lodotra, starting dose of 15mg administered in the evening
  Interventions: Drug: Lodotra®
- Prednisone IR (Active Comparator): Prednisone IR 15mg daily start dose (immediate release) administered in the morning
  Interventions: Drug: Prednisone IR (immediate release)

INTERVENTIONS:
Drug: Lodotra® — Lodotra, starting dose of 15mg administered in the evening
  Other Names: Modified release prednisone
  Arms: Lodotra®
Drug: Prednisone IR (immediate release) — Prednisone IR 15mg daily start dose (immediate release) administered in the morning,
  Arms: Prednisone IR

SUMMARY:
The study compares the efficacy and safety of modified release prednisone versus immediate release prednisone in patients suffering from polymyalgia rheumatica.

DETAILED DESCRIPTION:
The study consists of a screening phase, followed by a 4 week double-blind phase. During the double-blind phase, the patients will be randomised in a 1:1 ratio to either Lodotra® or immediate release prednisone (prednisone IR) plus respective placebo.

After completion of the double-blind phase, patients will be re-randomised in a 1:1 ratio to open-label Lodotra® or prednisone IR for 48 weeks. During the open-label phase, the dose of study medication will be tapered based on titration criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 50 years of age or older who provided written informed consent.
2. Females less than one year post-menopausal must have a negative serum or urine pregnancy test recorded prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner).
3. Subjects newly diagnosed with polymyalgia rheumatica and previously untreated with glucocorticoids for PMR. The diagnosis of polymyalgia rheumatica must be confirmed by all of the following criteria:

   * New onset bilateral shoulder pain or new onset bilateral shoulder and hip girdle pain.
   * PMR VAS score over the last 24 hours before the Screening Visit ≥ 50 (on a 0 - 100 scale).
   * Morning stiffness duration of ≥ 45 min on the day before the Screening Visit.
   * Acute phase response shown by elevated C-reactive protein (CRP; ≥ 2 times ULN).
4. Subjects willing and able to participate in all aspects of the study and comply with the use of study medication.

Exclusion Criteria:

1. Females who are pregnant (positive β-hCG test) or lactating.
2. Subjects with any contraindication/history of hypersensitivity to predniso(lo)ne or other ingredients.
3. Significant renal impairment (serume creatinine > 150 µmol/L).
4. Significant hepatic impairment (ALT, AST and GGT > 2.5 ULN).
5. Subjects suffering from another disease which requires glucocorticosteroid treatment. Topical glucocorticosteroids, e.g. intra-nasal or inhaled glucocorticosteroids are allowed but should be kept at a stable dose throughout the study.
6. Continued use of systemic glucocorticoids within 4 weeks prior to the Screening Visit.
7. Joint injections with glucocorticoids within 6 weeks prior to the Screening Visit.
8. Subjects who require treatment with non-permitted concomitant therapies.
9. Evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal or psychiatric disease at the time of screening, as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that would place the subject at risk upon exposure to the study medication or that may confound the analysis and/or interpretation of the study results.
10. Active alcohol or drug abuse.
11. Subjects suffering from giant cell arteritis, late onset rheumatoid arthritis or other inflammatory rheumatoid diseases.
12. Subjects suffering from drug-induced myalgia.
13. Subjects suffering from fibromyalgia
14. Subjects suffering from systemic lupus erythemathosus.
15. Subjects suffering from neurological conditions, e.g. Parkinson's disease.
16. Subjects suffering from active cancer.
17. Subjects suffering from an active infection.
18. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days prior to the Screening Visit.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To show that treatment with Lodotra® is noninferior to treatment with prednisone IR with regards to the percentage of complete responders. | 4 weeks

SECONDARY OUTCOMES:
Patient reported outcomes | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Southend University Hospital, Westcliff-on-Sea, United Kingdom

REFERENCES:
- See also: Link to Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=LOD3501